CLINICAL TRIAL: NCT05458856
Title: An Open-label, Multicentre, Single Arm Study to Assess the Efficacy and Safety of Triptorelin 6-month Formulation Administered Subcutaneously in Participants With Locally Advanced and/or Metastatic Prostate Cancer Previously Treated and Castrated With a GnRH Analogue
Brief Title: Effects of Triptorelin When Given Every 6-months Under the Skin to Adult Males With Cancer in the Prostate
Acronym: TriptoSwitch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-FR-52014-245; 2021-005719-29 (EudraCT Number)
Record Dates: First submitted 2022-06-17; First posted 2022-07-14 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Triptorelin embonate (Experimental): All participants will receive triptorelin embonate 22.5 mg
  Interventions: Drug: Triptorelin embonate 22.5 mg

INTERVENTIONS:
Drug: Triptorelin embonate 22.5 mg — A prolonged release formulation of triptorelin pamoate 22.5 mg 6-month formulation in D, L-lactide-co-glycolide polymers for single subcutaneous injection on Day 1 and Day 169
  Other Names: Decapeptyl

SUMMARY:
The aim of the study is to determine if triptorelin formulated for use every 6 months (given twice during the study) is effective and safe for when given by injection under the skin for the treatment of adult males with cancer in the prostate.

ELIGIBILITY:
Inclusion Criteria :

* Participant is male and must be 18 years of age inclusive, at the time of signing the informed consent
* Participant has histologically or cytologically proven prostate cancer with rising PSA after failed local therapy or metastatic disease, or requiring radiotherapy, and be a candidate for long-term (i.e. >1 year) androgen deprivation therapy
* Participant requires a GnRH analogue treatment for a minimum of 18 months, of which a minimum of 3 months of GnRH analogue treatment has already been provided prior to screening. (Note: participants must receive study intervention on Day 1 in accordance with the treatment schedule of their previously received GnRH analogue therapy).
* Has serum testosterone levels <1.735 nmol/L (50 ng/dL) at screening
* Has Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1
* Has a life expectancy of >18 months
* Male participants must agree that, if their partner is at risk of becoming pregnant (although highly unlikely in this study population), they will use an effective method of contraception. The participant must agree to use the contraception during the whole of the study and for 9 months after the last dose of study intervention
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol

Exclusion Criteria :

* Presence of another neoplastic lesion or brain metastases
* Metastatic hormone-sensitive prostate cancer with high tumour burden
* Metastatic castration-resistant prostate cancer
* Any concomitant disorder or resulting therapy that is likely to interfere with participant compliance or with the study in the opinion of the investigator
* Use of finasteride (Proscar®) or dutasteride (Avodart®/Avolve®) within the past 6 months
* Planned intermittent scheme of GnRH analogue
* At the time of screening, planned use of any chemotherapy for prostate cancer during the study
* Prior hypophysectomy or adrenalectomy
* Participation in another study with an experimental drug within 3 months before signing informed consent or within five half-lives of the investigational drug (whichever was the longer), or any other type of medical research
* Severe kidney or liver failure (creatinine >2 times the normal range, aspartate aminotransferase and alanine aminotransferase >3 times the normal range)
* Any concomitant disorder or resulting therapy that is likely to interfere with participant's compliance, the subcutaneous administration of the drug or with the study in the opinion of the investigator
* Previous history of QT prolongation or concomitant use of medicinal products known to prolong the QT interval or with a known risk of torsades de pointes
* Known hypersensitivity to triptorelin or any of its excipients, GnRH, other GnRH agonist/analogues
* Known active use of recreational drug or alcohol dependence in the opinion of the investigator
* Inability to give informed consent or to comply fully with the protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant is male as indication is prostate cancer
Enrollment: 147 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (39):
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Antwerpen, Edegem
  - AZGroeninge, Kortrijk
  - CHU de Liège - Domaine Universitaire du Sart Tilman - Urologie, Liège
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- France (11):
  - Centre Hospitalier Universitaire D'Angers - Urologie, Angers
  - CHU Brest-Hopital Morvan Institut de Cancerologie et d'Hemat, Brest
  - Clinique Pasteur-Lanroze - Oncology, Brest
  - Polyclinique de Blois - Service oncologie, La Chaussée-Saint-Victor
  - Hopital Privé Métropole Lille - Polyclinique Du Bois, Lille
  - CHU Hopital Edouard Herriot, Lyon
  - L'Institut Mutualiste Montsouris, Paris
  - Hopital Bichat, Paris
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Foch - Urologie et Transplantation Ré, Suresnes
  - Saint Jean Languedoc and La Croix du Sud Hospital, Toulouse
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - University Hospital Jena KöR, Jena
  - Universitaetsklinikum Muenster, Münster
  - Studienpraxis Urologie, Nürtingen
  - Universität Tuebingen - Urology, Tübingen
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - National Cancer Institute, Vilnius
  - Vilniaus Universiteto ligonines Santariskiu Klinikos, Vilnius
- Netherlands (4):
  - The Netherlands Cancer Institute - Oncology, Amsterdam
  - Catharina Ziekenhuis - Urology, Eindhoven
  - CWZ, Nijmegen
  - Haga Ziekenhuis, The Hague
- Spain (8):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de La Santa Creu i Sant Pau - Oncología Médica, Barcelona
  - H. de Basurto - Urología, Bilbao
  - POLUSA - Policlínico Lucense - Oncología, Lugo
  - Hospital Universitario 12 de Octubre- Urology, Madrid
  - Hospital Universitario Central de Asturias (HUCA), Oviedo
  - Hospital Universitario Virgen del Rocio- Urología Pediátrica, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2025/07/04145025/D-FR-52014-245_Lay-Summary_Final_04Jul2025.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, multicenter, open-label, single arm study was conducted at 26 investigational sites in 6 countries from 30-Aug-2022 to 08-Jul-2024 in participants with locally advanced and/or metastatic prostate cancer previously treated and castrated with a gonadotropin-releasing hormone (GnRH) analogue.
Pre-assignment Details: The study consisted of a screening period (Day -28 to Day -1), study treatment administration on Days 1 and 169 (with visits on Days 3, 7, 29, 85, 141, 171, 175, 253, 309) and an end of study/early discontinuation visit on Day 337. A total of 147 participants were enrolled in the study.
Groups:
- Triptorelin Embonate 22.5 mg: Participants received triptorelin embonate 22.5 milligrams (mg) subcutaneous (SC) injection on Days 1 and 169.
Period: Overall Study
Arm/Group | Triptorelin Embonate 22.5 mg
Started | 147
Received Treatment | 145
Completed | 134
Not Completed | 13
Not completed — Withdrawal by Subject | 5
Not completed — Death | 4
Not completed — Protocol Deviation | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The enrolled set included all participants who were enrolled to study treatment.
Groups:
- Triptorelin Embonate 22.5 mg: Participants received triptorelin embonate 22.5 mg SC injection on Days 1 and 169.
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 104
  Unknown or Not Reported | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 109
  Other | 2
  Not Reported | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintained Castrate Levels of Serum Testosterone During the Study
Description: Blood samples were collected for the measurement of serum testosterone concentrations using a validated, specific and sensitive liquid chromatography tandem mass spectrometry method. Maintenance of castration during the study was defined as testosterone <1.735 nanomoles per liter (nmol/L) (<50 nanograms/deciliter [ng/dL]) at Days 29, 85, 141, 169, 253, 309 and 337.
Time Frame: Up to Day 337
Population: The full analysis set (FAS) included all participants who signed an informed consent form (ICF) and received 2 administrations of study treatment and completed all visits for testosterone measurement (Days 29, 85, 141, 169, 253, 309 and 337).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 120
percentage of participants | 95.0 [89.4 to 98.1]

2. Secondary Outcome: Percentage of Participants Castrated on Days 29, 85, 141, 169, 253, 309 and 337
Description: Blood samples were collected for the measurement of serum testosterone concentrations using a validated, specific and sensitive liquid chromatography tandem mass spectrometry method. Castration was defined as testosterone <1.735 nmol/L (<50 ng/dL).
Time Frame: Days 29, 85, 141, 169, 253, 309 and 337
Population: The FAS included all participants who signed an ICF and received 2 administrations of study treatment and completed all visits for testosterone measurement (Days 29, 85, 141, 169, 253, 309 and 337).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 120
percentage of participants
  Day 29 | 100.0 [97.0 to 100.0]
  Day 85 | 100.0 [97.0 to 100.0]
  Day 141 | 98.3 [94.1 to 99.8]
  Day 169 | 97.5 [92.9 to 99.5]
  Day 253 | 100.0 [97.0 to 100.0]
  Day 309 | 99.2 [95.4 to 100.0]
  Day 337 | 99.2 [95.4 to 100.0]

3. Secondary Outcome: Percentage of Participants With a Serum Testosterone Level <0.694 Nmol/L (<20 ng/dL) During the Study
Description: Blood samples were collected for the measurement of serum testosterone concentrations using a validated, specific and sensitive liquid chromatography tandem mass spectrometry method.
Time Frame: Up to Day 337
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 120
percentage of participants | 83.3 [75.4 to 89.5]

4. Secondary Outcome: Percentage of Participants With a Serum Testosterone Level <0.694 Nmol/L (<20 ng/dL) on Days 29, 85, 141, 169, 253, 309 and 337
Description: as for outcome 3
Time Frame: Days 29, 85, 141, 169, 253, 309 and 337
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 120
percentage of participants
  Day 29 | 92.5 [86.2 to 96.5]
  Day 85 | 92.5 [86.2 to 96.5]
  Day 141 | 92.5 [86.2 to 96.5]
  Day 169 | 94.2 [88.4 to 97.6]
  Day 253 | 95.8 [90.5 to 98.6]
  Day 309 | 95.8 [90.5 to 98.6]
  Day 337 | 98.3 [94.1 to 99.8]

5. Secondary Outcome: Percentage of Participants Castrated on Days 3 and 7 After Each Injection Administered on Days 1 and 169
Description: as for outcome 2
Time Frame: On Days 3, 7, 171, and 175
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 120
percentage of participants
  Day 3 | 92.5 [86.2 to 96.5]
  Day 7 | 98.3 [94.1 to 99.8]
  Day 171 | 95.0 [89.4 to 98.1]
  Day 175 | 95.8 [90.5 to 98.6]

6. Secondary Outcome: Percent Change From Baseline in Prostate Specific Antigen (PSA) at Days 169 and 337
Description: Blood samples were collected for the measurement of plasma PSA concentrations. Percent change in PSA was defined as the absolute value of the difference between the PSA values at Days 169 and 337 and the baseline value divided by the baseline value. The baseline value was the last sample prior to the first injection.
Time Frame: Baseline (prior to injection on Day 1), Days 169 and 337
Population: The FAS included all participants who signed an ICF and received 2 administrations of study treatment and completed all visits for testosterone measurement (Days 29, 85, 141, 169, 253, 309 and 337). Only those participants with data collected at specified timepoints are reported.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 118
percent change
  Day 169: number analyzed (Participants) | 115
  Day 169 | 0.00 [-35.60 to 0.00]
  Day 337 | 0.00 [-46.90 to 14.30]

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and TEAEs of Local Intolerance
Description: An adverse event (AE) was any untoward medical occurrence in clinical study participant, temporally associated with use of study treatment, whether or not considered related to study treatment. TEAEs were AEs that started or worsened on or after the first study treatment administration and within 168 days after the last dose of study treatment, or up to Day 337, whichever was later. Local tolerance was assessed 2 hours after each injection by examination of injection site for signs such as but not limited to tenderness, redness, bruising, erythema, swelling, rash, pain, itching, induration, hematoma, ulceration or necrosis.
Time Frame: From first dose of study treatment (Day 1) up to end of study visit (Day 337)
Population: The safety set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 145
Participants
  TEAEs | 88
  TEAEs of Local Intolerance | 19

ADVERSE EVENTS:
Time Frame: Serious AEs, non-serious AEs and all-cause mortality (deaths) were collected from screening (Day -28) up to end of study visit (Day 337), up to maximum of 365 days
Description: The safety set included all participants who received at least 1 dose of study treatment.
Arm/Group | Triptorelin Embonate 22.5 mg
All-Cause Mortality (participants affected / at risk) | 4/145
Serious Adverse Events (participants affected / at risk) | 26/145
Other Adverse Events (participants affected / at risk) | 38/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Embonate 22.5 mg (N=145)
COVID-19 (Infections and infestations) | 4 (4)
Anal abscess (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Peroneal nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Disease progression (General disorders) | 2 (2)
Death (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Embonate 22.5 mg (N=145)
Hot flush (Vascular disorders) | 17 (18)
Hypertension (Vascular disorders) | 14 (15)
Fall (Injury, poisoning and procedural complications) | 9 (9)
Fatigue (General disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT05458856/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT05458856/SAP_001.pdf